CLINICAL TRIAL: NCT05406479
Title: Bedaquiline Enhanced Post ExpOsure Prophylaxis for Leprosy: Phase 2 Study
Brief Title: Bedaquiline Enhanced Post ExpOsure Prophylaxis for Leprosy (Phase 2)
Acronym: BE-PEOPLE P2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Damien Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BE-PEOPLE Phase 2
Record Dates: First submitted 2022-05-20; First posted 2022-06-06 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy | interventions — bedaquiline; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BE-PEP (Bedaquiline Post-Exposure Prophylaxis) (Experimental): Eligible participants will receive one dose of Bedaquiline plus Rifampicin
  Interventions: Drug: BE-PEP (Bedaquiline); Drug: BE-PEP (Rifampicine)
- SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis) (Active Comparator): Eligible participants will receive one dose of Rifampicin (WHO recommendation)
  Interventions: Drug: SDR-PEP

INTERVENTIONS:
Drug: BE-PEP (Bedaquiline) — Single dose of Bedaquiline
  Arms: BE-PEP (Bedaquiline Post-Exposure Prophylaxis)
Drug: SDR-PEP — Single dose of Rifampicin
  Arms: SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis)
Drug: BE-PEP (Rifampicine) — Single dose of Rifampicin
  Arms: BE-PEP (Bedaquiline Post-Exposure Prophylaxis)

SUMMARY:
This study will evaluate a combination of bedaquiline and rifampicin as post exposure prophylaxis (PEP) for leprosy in Comoros. It will be a follow-up to the PEOPLE trial on PEP with rifampicin, which is ending in 2022. This new trial will be called the 'Bedaquiline Enhanced Post ExpOsure Prophylaxis for Leprosy' or 'BE-PEOPLE' trial. There will be two main study arms, a comparator arm based on the current WHO recommendation of providing a single dose of rifampicin (10 mg/kg) to close contacts of leprosy patients and an intervention arm in which this regimen will be reinforced with bedaquiline, 400 or 800 mg depending on weight, to be repeated once after four weeks for household contacts. The main study will be preceded by a phase 2 safety study.

DETAILED DESCRIPTION:
Given the fact that the investigators are going to provide to healthy people a drug that has not been used before for this indication and which has only been conditionally approved for use in multi-drug resistant tuberculosis, they have first foreseen a phase 2 study in which BE-PEP will be provided to a limited number of contacts and in which safety will be closely monitored and evaluated by an independent data and safety monitoring board (DSMB). This will be done in a small village that is part arm 1 of the PEOPLE trial in which 8 new cases have been diagnosed since 2019 but no PEP has been provided. The investigators will conduct door-to-door screening in this village in June 2022 and offer a single dose of BE-PEP to a random sample of 150 people screened aged 5 years and above not meeting the exclusion criteria (active tuberculosis (TB) or leprosy or previously treated leprosy, known liver function or cardiac abnormalities, not able to swallow 100 mg bedaquiline tablets). Participants will be followed up closely with active monitoring for adverse events, including measurement of the corrected QT interval and liver function before and after administration, as well as gastro-intestinal (nausea, vomiting), nervous system-related (headache, dizziness) and cutaneous reactions. The remainder of the population of this village aged two years and above will be offered single dose rifampicin as per WHO recommendations. In a randomly sampled subset of 150 individuals receiving rifampicin only, the same stringent monitoring with ECG and liver function tests also applied in those receiving BE-PEP will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Being a permanent resident of the study village, in good state of health
2. Able and willing to provide informed consent
3. Age 5 years or above and weight of 20 kg or above

Exclusion Criteria:

1. Signs of active leprosy
2. Signs of active pulmonary tuberculosis (cough ≥2 weeks duration)
3. Signs of active extra-pulmonary tuberculosis (bluish-red nodules that cover the lymph nodes, bones or joints, or cervical glands with discharge)
4. History of liver- or kidney disease
5. Allergy to rifampicin or bedaquiline
6. Having received rifampicin or bedaquiline (if applicable) in the last 2-year period
7. Not able to swallow bedaquiline 100 mg tablets
8. Self-reported (suspected) pregnancy or breastfeeding
9. Concurrent (within the last three week period before D0) use of medications not included in the safe list (for bedaquiline only)
10. QT-prolongation of ≥450 msec in baseline ECG within the last week.
11. Jaundice or self-reported liver function abnormalities or hepatitis
12. Value of baseline ALT or AST >3x ULN within the last week. In case only ALT is available, this would suffice for enrollment

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Younoussa Assoumani, Principal Investigator — Damien Foundation Comoros
Locations (1):
- Fondation Damien, Gege, Ndzuwani, Comoros

REFERENCES:
- [Derived] de Jong BC, Nourdine S, Bergeman AT, Salim Z, Grillone SH, Braet SM, Wirdane Abdou M, Snijders R, Ronse M, Hoof C, Tsoumanis A, Ortuno-Gutierrez N, der Werf CV, Piubello A, Mzembaba A, Assoumani Y, Hasker E. Safety of single-dose bedaquiline combined with rifampicin for leprosy post-exposure prophylaxis: A Phase 2 randomized non-inferiority trial in the Comoros Islands. PLoS Med. 2024 Oct 21;21(10):e1004453. doi: 10.1371/journal.pmed.1004453. eCollection 2024 Oct. PMID 39432509

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis)
Started | 157 | 156
Completed | 156 | 154
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis) | Total
Number analyzed (Participants) | 157 | 156 | 313
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 62 | 126
  Between 18 and 65 years | 93 | 94 | 187
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [31 to 53] | 41 [32 to 54.5] | 41 [32 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 83 | 167
  Male | 73 | 73 | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Comoros | 157 | 156 | 313

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in QTc Interval Between the Two Arms 24 Hours After Treatment Administration
Description: Mean difference in QTc interval between the two arms 24 hours after treatment administration.
  Difference (BE-PEP - SDR-PEP)
Time Frame: 24 hours after treatment administration
Population: participants included per protocol
Measure: Mean (95% Confidence Interval); unit: msec
Groups:
- BE-PEP (Bedaquiline Post-Exposure Prophylaxis): Participants received bedaquiline and rifampicine as PEP treatment
- SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis): Participants received rifampicine as PEP treatment
Arm/Group | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis)
Number analyzed (Participants) | 150 | 146
msec
  Adults (> 18): number analyzed (Participants) | 88 | 85
  Adults (> 18) | 396.81 [392.45 to 401.17] | 397 [392.94 to 401.06]
  Adolescents (13 - 17): number analyzed (Participants) | 18 | 18
  Adolescents (13 - 17) | 404.61 [395.43 to 413.79] | 394.06 [386.33 to 401.79]
  Children (5 - 12): number analyzed (Participants) | 44 | 43
  Children (5 - 12) | 391.15 [386.36 to 395.94] | 389.07 [384.52 to 393.62]
Statistical Analysis 1: Comparison: BE-PEP (Bedaquiline Post-Exposure Prophylaxis) vs SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis); Adults; Test type: Non-Inferiority — For the hypothesis testing of non-inferiority the confidence interval should be compared to the non-inferiority margin. More specifically, non-inferiority is established if the upper limit of a one-sided 95% confidence interval around the difference in means QTc 24 hours after treatment administration (BE-PEP - SDR-PEP) is below the non-inferiority limit of +10 ms. A two-sample t-test was used to compare the two groups, but the p-value returned should not be used to conclude non-inferiority; Mean Difference (Final Values) = -0.193, 95% CI 2-sided [-5.146 to 4.76]
Statistical Analysis 2: Comparison: BE-PEP (Bedaquiline Post-Exposure Prophylaxis) vs SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis); Adolescents (13-17); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.556, 95% CI 2-sided [0.926 to 20.185]
Statistical Analysis 3: Comparison: BE-PEP (Bedaquiline Post-Exposure Prophylaxis) vs SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis); Children (5-12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.076, 95% CI 2-sided [-3.374 to 7.525]

2. Primary Outcome: Occurence of Any Predetermined Study Stopping Criteria, Which Will Trigger an Immediate Pause on Enrollment
Description: Occurence of any of the following predetermined study stopping criteria, which will trigger an immediate pause on enrollment:
  1. Death of a participant considered related to study drug
  2. One or more participants experience an Serious Adverse Event (SAE) or Grade 4 Adverse Event (AE) or a persistent (upon repeat testing) Grade 4 laboratory abnormality that is determined to be related to study drug
  3. Three or more participants experience a Grade 3 or greater AE of the same type (as per medical judgement) that is determined to be related to study drug
  4. Three or more participants experience a persistent (upon repeat testing) Grade 3 laboratory abnormality related to the same laboratory parameter and considered to be related to study drug
  5. Two or more participants experience QTc > 500 ms
  6. One or more participants has Aspartate transaminase (AST) or Alanine transaminase (ALT) > 8x Upper limit of normal (ULN), in absence of causative explanation
Time Frame: Until day 30 after treatment administration
Population: included in per protocol
Measure: Count of Participants; unit: Participants
Groups:
- BE-PEP (Bedaquiline Post-Exposure Prophylaxis): received bedaquiline and rifampicine as PEP treatment
- SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis): received rifampicine as PEP treatment
Arm/Group | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis)
Number analyzed (Participants) | 157 | 156
Participants
  Adults (> 18): number analyzed (Participants) | 93 | 94
  Adults (> 18) | 0 | 0
  Adolescents (13 - 17): number analyzed (Participants) | 20 | 18
  Adolescents (13 - 17) | 0 | 0
  Children (5 - 12): number analyzed (Participants) | 44 | 44
  Children (5 - 12) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected between administration of the medication (day 1 of the study) until 30 days post administration
Arm/Group | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/156
Serious Adverse Events (participants affected / at risk) | 1/157 | 1/156
Other Adverse Events (participants affected / at risk) | 65/157 | 50/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) (N=157) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis) (N=156)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BE-PEP (Bedaquiline Post-Exposure Prophylaxis) (N=157) | SDR-PEP (Single-Dose Rifampicin Post-Exposure Prophylaxis) (N=156)
Palpitations (Cardiac disorders) | 4 | 1
Vertigo (Ear and labyrinth disorders) | 14 | 10
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 13 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 0 | 1
malaise (General disorders) | 1 | 0
pyrexia (General disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 14 | 22
Aspartate aminotransferase increased (Investigations) | 22 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 17 | 2
Tremor (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05406479/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT05406479/SAP_001.pdf